CLINICAL TRIAL: NCT03758495
Title: Rescuing the Ruminating Brain: Identifying Biomarkers of Rumination and Mindfulness Through Concurrent EEG and fMRI Studies of Schizophrenia and Depression
Brief Title: Rescuing the Ruminating Brain: Identifying Biomarkers of Rumination and Mindfulness Through Concurrent EEG and Functional Magnetic Resonance Imaging (fMRI) Studies of Schizophrenia and Depression
Status: Withdrawn | Type: Observational
Why Stopped: This study was not intended to be published as a trial.
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: MHBB-012-17S; CX000497 (Other Grant/Funding Number: eRA Project Reference)
Record Dates: First submitted 2018-11-07; First posted 2018-11-29 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Schizophrenia; Depressive Disorder, Major
MeSH Terms: conditions — Schizophrenia; Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Patients with Schizophrenia: Individuals who have been previously diagnosed with schizophrenia and meet our research criteria for symptoms indicative of schizophrenia within their lifetime.
  Interventions: Other: Electroencephalography (EEG) and Magnetic Resonance Imaging (MRI)
- Patients with Major Depressive Disorder: Individuals who have been previously diagnosed with major depressive disorder and meet our research criteria for symptoms indicative of major depressive disorder within their lifetime.
  Interventions: Other: Electroencephalography (EEG) and Magnetic Resonance Imaging (MRI)
- Healthy Controls: Individuals who have not met criteria for a psychiatric disorder within their lifetime according to our research criteria for symptoms indicative of a psychiatric disorder.
  Interventions: Other: Electroencephalography (EEG) and Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Other: Electroencephalography (EEG) and Magnetic Resonance Imaging (MRI) — The investigators will use these techniques combined with attention tests, memory tests, and clinical interviews to explore connections between these measures and activity in the brain in patients with a diagnosis of schizophrenia, major depressive disorder, and healthy controls.

SUMMARY:
The investigators will acquire simultaneous EEG and fMRI data from Veterans with depression and schizophrenia and mentally healthy Veterans to assess early sensory responses, context updating, and responses to emotional images. Understanding how rumination affects engagement with the environment is the first step towards assessing its far-reaching cognitive and emotional costs, which cut across traditional diagnostic boundaries. Understanding how mindfulness restores information processing will increase our understanding of how, and for whom, it works.

DETAILED DESCRIPTION:
Is "the idle mind the devil's playground?" It depends on where the wandering mind goes. If it is busy reflecting on recent activity, consolidating recent material into long term memories, and envisioning the future, then these thought patterns may be highly adaptive, allowing us to learn from the past and plan for the future. But when the mind turns to the dark side and rumination takes over, these thought patterns are maladaptive. Rumination involves recursive negative thinking focused on causes and consequences rather than solutions. It cuts across diagnostic boundaries: it is both a cause and consequence of major depressive disorder (MDD) and is related to hallucinations and delusions in schizophrenia (SZ). It affects cognitive and emotional responses, yet it can be treated with mindfulness-based therapies.

Mindfulness-meditation is a type of behavioral therapy that focuses on cultivating present focused attention, is a stress-reduction intervention that targets rumination, and improves many medical and psychiatric conditions: Trait mindfulness is associated with less distress from auditory hallucinations and fewer residual depressive symptoms. It is the practice of attending to present moment experiences and allowing emotions and thoughts to come and go without judgment, thereby avoiding a downward spiral into rumination.

Compared to simple mind wandering, a brief mindfulness induction recruits an attention network including parietal and prefrontal structures while mind wandering only recruits the default mode network (DMN) Based on data from the last funding period, the investigators know that activation of the DMN affects both basic sensory and semantic processing in SZ. The investigators propose to extend this by focusing specifically on rumination and adding patients with depression. The investigators ask how rumination affects basic sensory, cognitive and emotional responses, and if mindfulness can rescue these functions, across diagnoses and the wellness spectrum.

The investigators will acquire simultaneous EEG and fMRI data from Veterans with depression and schizophrenia and mentally healthy Veterans to assess early sensory responses, context updating, and responses to emotional images. Understanding how rumination affects engagement with the environment is the first step towards assessing its far-reaching cognitive and emotional costs, which cut across traditional diagnostic boundaries. Understanding how mindfulness restores information processing will increase our understanding of how, and for whom, it works.

The investigators predict rumination inductions will prevent the brain from fully processing a spectrum of external events, and mindfulness inductions will restore these abilities. The investigators predict trait rumination and mindfulness will modulate the effects in all groups, with exaggerated effects in those with depression or schizophrenia. The outcome variables will be EEG-based event related potentials (ERPs) and fMRI, and their integration. Symptom severity, trait rumination, and trait mindfulness will be considered in the analyses.

Aim 1: Simple effects of rumination inductions on fMRI connectivity. The investigators will compare the effects of rumination and mindfulness inductions on the connectivity between DMN and rumination-sensitive brain regions. Compared to mindfulness inductions, the investigators predict rumination will increase this connectivity, with greater effects in depressed and schizophrenia patients than in healthy controls.

Aim 2: Carry-over effects of mindfulness inductions on ERPs and fMRI and their integration. The investigators predict the effects of 30-second mindfulness inductions will persist into the subsequent visual oddball task, thereby augmenting sensory, attention, and emotional ERP components and fMRI activation in sensory, cognitive and emotional networks, compared to rumination inductions. The investigators will explore the covariance between fMRI and ERP data fusion methods as they have done previously.

Aim 3: Effects of trait rumination and mindfulness. The investigators will assess the relationship between neural data and trait rumination, mindfulness, and symptom severity in all groups.

ELIGIBILITY:
Inclusion Criteria:

(All)

* Veterans
* 18-65 years of age
* Negative metal screen for MR scanning
* Corrected to normal vision

Inclusion Criteria (patients):

* Meet criteria for SZ or MDD as assessed using the Structured Clinical Interview for DSM (SCID), with a consensus diagnosis between trained research staff member and an attending psychiatrist or psychologist.
* Stable medication regime for > 1 month

Exclusion Criteria:

(All)

* Past or present neurological problems (including seizures and head trauma resulting in neurological or cognitive sequelae)
* Loss of consciousness (LOC) greater than 30 minutes or any LOC with neurologic sequelae
* Major medical conditions (e.g., significant hypertension, diabetes not controlled by diet alone, seizure disorders, treatment with anticonvulsant medication, endocrine disorders, significant cardiac pathology)
* Substance abuse within three months of participation or any history of substance dependence
* History of HIV risk behaviors
* Known claustrophobia
* Pregnancy. If the participant cannot rule out pregnancy, a pregnancy urine test will be conducted moments before scanning.
* Uncorrected vision as assessed by the Snellen chart.

Exclusion criteria (patients only):

- Any primary Diagnostic and Statistical Manual Diploma in Social Medicine (DSM) Axis I diagnosis other than SZ or MDD

Exclusion criteria (controls only):

* Any past or present DSM Axis I diagnosis
* Chronic treatment with medication that affects cognitive function

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have been diagnosed with schizophrenia and meet our research criteria of symptoms indicative of a diagnosis of schizophrenia within their lifetime are eligible for this study.
  Patients who have been diagnosed with major depressive disorder and meet our research criteria of symptoms indicative of a diagnosis of major depressive disorder within their lifetime are eligible for this study.
  Healthy controls who have never met criteria for a psychiatric disorder and meet our research criteria will also be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2018-11-02 (Actual)

PRIMARY OUTCOMES:
Electroencephalography (EEG) | Day 1
  Electroencephalography, measures signals from the brain while participants conduct specific tasks that measure memory and attention.
Magnetic Resonance Imaging (MRI) | Day 1
  Magnetic Resonance Imaging, measures activity in, and takes detailed pictures of the brain while participants conduct specific tasks that measure memory and attention.
Memory and Attention task | Day 1
  Listening to audio instructions.

CONTACTS AND LOCATIONS:
Overall Officials: Judith M Ford, PhD, Principal Investigator — San Francisco VA Medical Center, San Francisco, CA
Locations (1):
- San Francisco VA Medical Center, San Francisco, CA, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No